CLINICAL TRIAL: NCT06196086
Title: Evaluation of Myocardial Stiffness in Patients With Heart Failure With Preserved Ejection Fraction by Intrinsic Wave Velocity Propagation
Brief Title: Myocardial Stiffness Evaluation in Patients With Heart Failure With Preserved Ejection Fraction
Status: Recruiting | Type: Observational
Sponsor: Haiyan Wang (Other)
Responsible Party: Sponsor-Investigator, Haiyan Wang, Director, Qianfoshan Hospital
Organization: Qianfoshan Hospital (Other)
Other Study IDs: YXLL-KY-2023（152）
Record Dates: First submitted 2023-12-23; First posted 2024-01-09 (Actual); Last update posted 2024-01-09 (Actual); Status verified 2024-01

CONDITIONS: Heart Failure With Preserved Ejection Fraction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- HFpEF: Patients who diagnosed with heart failure with preserved ejection fraction based on symptoms, serum biomarker and test according to 2022 AHA/ACC/HFSA Guidelines for Heart Failure Management at the First Affiliated Hospital of Shandong First Medical University from December 20, 2023 to December 20, 2026.
  Interventions: Diagnostic Test: Echocardiography examination
- Control: Healthy volunteers with no history of heart disease who matched for age, sex, and risk factors with HFpEF group.
  Interventions: Diagnostic Test: Echocardiography examination

INTERVENTIONS:
Diagnostic Test: Echocardiography examination — Echocardiography examination and software post-processing analysis was performed to obtain parameters of conventional echocardiography, left atrial and left ventricle strain, and IVP.

SUMMARY:
The goal of this observational study is to evaluating myocardial stiffness in patients with heart failure with preserved ejection fraction (HFpEF) by intrinsic wave velocity propagation (IVP). The main questions it aims to answer are:

* Whether myocardial stiffness assessed by IVP in patients with HFpEF Increased.
* Whether IVP is related to the cardiac structure and function in patients with HFpEF.
* What are the risk factors that may be associated with heart failure rehospitalization in patients with HFpEF?
* Whether increased myocardial stiffness is a risk factor for heart failure rehospitalization.

Participants will undergo transthoracic echocardiography to obtain conventional ultrasound parameters, and software post-processing analysis to obtained two-dimensional strain parameters and IVP, as well as general clinical data and laboratory test results. Clinical followed up was performed through electronic medical records or telephone interviews until patient rehospitalization for heart failure or discharge for one year.

DETAILED DESCRIPTION:
The included patients who diagnosed with HFpEF and healthy volunteers at the First Affiliated Hospital of Shandong First Medical University from December 20, 2023 to December 20, 2026. Routine clinical and echocardiographic data, two-dimensional strain parameters and IVP of the study subjects were obtained:

1. The echocardiographic examination was performed using a GE Vivid E95 ultrasound machine, and images were acquired with the patient in left lateral decubitus using a 3.5-5 MHz transducer at a depth of 16 cm. ECG was recorded, and 3 consecutive cardiac cycles of each view were recorded during quiet breathing at 50-80 frames/sec. All patients were subjected to conventional transthoracic echocardiography, Speckle tracking echocardiography and IVP. All measurements were taken following the American Society of Echocardiography (ASE) recommendations.
2. Left atrial and left ventricle strain analysis was obtained using automated speckle tracking software. The regions of interest were generated automatically and left atrial endocardial border was manually adjusted when required. Left atrial phases definition and left atrial strain values were measured from the Left atrial longitudinal strain curve according to the European Association of Cardiovascular Imaging (EACVI)/American society of echocardiography (ASE) guidelines. Global left ventricle strain was evaluated, and the software automatically traced the contour of the endocardium at apical three, four and two-chamber views.
3. For IVP analysis, we first entered Q-analysis and then used the curved anatomic M-mode to trace the left ventricle myocardium to reconstruct the axial tissue velocity maps. The tissue velocity map scale was adjusted to create velocity aliasing to better illustrate the is velocity wave front that propagated in the myocardium during end-diastole induced by atrial contraction. Sweep speed was adjusted to maximum, and the slope of the is velocity wave was measured as the propagation speed of the intrinsic wave. The average wave velocity was calculated using all measurements from all six myocardial walls using the three apical views.
4. At the same time, the general clinical data, demographic characteristics, electrocardiogram, coronary artery CTA, carotid ultrasound, and laboratory results include brain natriuretic peptide (BNP), uric acid (UA), soluble growth stimulating expression gene 2 protein (sST2), growth differentiation factor 15(GDF-15), Galectin-3 (Galectin-3) were obtained through electronic health record.
5. Clinical follow-up was performed every 6 months after discharge by phone and by electronic health record review until heart failure readmission or one year after discharge. Heart failure rehospitalization was defined as any rehospitalization during which HF was listed as one primary diagnosis based on typical heart failure symptoms, signs and increased B-type natriuretic peptide levels for which intravenous diuretics or increased dose of loop diuretics were needed in clinic.

ELIGIBILITY:
Inclusion Criteria:

Meet the diagnostic criteria for HFpEF in the 2022 AHA/ACC/HFSA Guidelines for Heart Failure Management:

* Present with signs and symptoms of heart failure;
* LVEF≥50%;
* There is at least one additional criterion: Increased BNP (BNP≥35pg/ml, NT-pro BNP>125pg/ml) and resting echocardiography measured E/e' ≥ 15; Stress echocardiography determined E/e' ≥ 15; Cardiac catheterization at rest, PCWP ≥ 15 mmHg or LVEDP ≥ 16 mmHg; The PCWP at peak exercise was ≥ 25 mmHg.

Exclusion Criteria:

* Acute coronary syndrome, acute heart failure or coronary revascularization in three months;
* HFimpEF, cardiomyopathy, severe valvular heart disease, arrhythmia;
* Thyroid dysfunction, pulmonary hypertension, past or current pulmonary embolism, severe chronic obstructive pulmonary disease, malignancy/renal failure (less than 30) ml/min);
* Poor echocardiogram image quality.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients who diagnosed with HFpEF according to the 2022 AHA/ACC/HFSA Guidelines for Heart Failure Management.
Sampling Method: Non-Probability Sample
Enrollment: 438 (Estimated)
Dates: Start 2023-12-20 (Actual); Primary Completion 2026-12-20 (Estimated); Study Completion 2027-12-20 (Estimated)

PRIMARY OUTCOMES:
IVP | After recruiting, IVP collected through software post-processing analysis will be assessed and reported up to 8 weeks.
  The propagating wave velocity along longitudinal tissue motion direction is referred to as the Intrinsic Velocity Propagation (IVP). It is generated through the dynamic nature of the heart and allows quantification in all LV segments. It is possible that this wave is related to tissue stiffness and has a radial component.

CONTACTS AND LOCATIONS:
Overall Officials: Haiyan Wang, Principal Investigator — Shandong First Medical University
Locations (1):
- The First Affiliated Hospital of Shandong First Medical University, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: No